CLINICAL TRIAL: NCT02629146
Title: A Single Center, Prospective, Randomized, Double Blind, Placebo-controlled, Three-way Cross-over Study of the Analgesic Effects of Midazolam Versus Placebo With Fentanyl as an Active Control in Human Volunteers
Brief Title: Analgesic Effects of Midazolam in Human Volunteers
Acronym: GabA01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Akron Molecules AG (Industry)
Responsible Party: Principal Investigator, Burkhard Gustorff, Univ.Prof. Dr., Wilhelminenspital Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GabA01
Record Dates: First submitted 2015-12-06; First posted 2015-12-14 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Analgesic Drugs; Antinociceptive Agents
Keywords: Midazolam; Fentanyl
MeSH Terms: interventions — Midazolam; Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midazolam (Experimental): Drug: Midazolam (experimental)
  Interventions: Drug: Midazolam
- Isotonic saline (Placebo Comparator): Drug: Isotonic saline (placebo)
  Interventions: Drug: Isotonic saline
- Fentanyl (Active Comparator): Drug: Fentanyl (active comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Midazolam
  Other Names: Dormicum
  Arms: Midazolam
Drug: Fentanyl
  Arms: Fentanyl
Drug: Isotonic saline
  Arms: Isotonic saline

SUMMARY:
This study evaluates analgesic properties of midazolam compared to placebo and fentanyl. Each participant will receive all three drugs (midazolam, fentanyl, placebo) on three different occasions (study visits) and the effect on different pain stimuli will be tested.

ELIGIBILITY:
Inclusion Criteria:

* male and female volunteers
* 18-40 years old
* healthy
* body mass index between 5th and 85th percentile
* Caucasian
* non smoker or moderate smoker (<10 cigarettes per day)
* able to understand, write, and read German

Exclusion Criteria:

* acute or chronic pain condition (except for mild day-to-day pain on <5 days/month)
* previous (up to 5 days preceding the study) or current medications prescription or over-the-counter, especially analgesics
* symptoms of a clinically relevant illness in the 2 weeks before the first study day
* hypertension
* any known psychiatric condition
* abuse of alcoholic beverages, drug abuse
* known positive human immunodeficiency virus status
* any known medical condition which may interact with study medication, study objectives, or compliance of subject with study tasks
* participation in a clinical trial in the 4 weeks preceding the study
* known allergy against Midazolam
* known allergy against Fentanyl
* pregnancy or breast-feeding
* unable or unwilling to give informed consent
* unable or unwilling to follow investigator's instructions
* unable or unwilling to comply with study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in pain ratings (0-100) to a suprathreshold heat pain stimulus | 3.5 Minutes after end of infusion

SECONDARY OUTCOMES:
Change in pain ratings to a suprathreshold electrical pain stimulus | 3.5 Minutes after end of infusion
Increase of pressure pain thresholds (kPa) | Up until 23 Minutes after end of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Gustorff, Prof.Dr., Principal Investigator — Wilhelminenspital Vienna
Locations (1):
- Schmerzdiagnostik / Clinical Research Unit, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laursen DR, Nejstgaard CH, Bjorkedal E, Frost AD, Hansen MR, Paludan-Muller AS, Prosenz J, Werner CP, Hrobjartsson A. Impact of active placebo controls on estimated drug effects in randomised trials: a systematic review of trials with both active placebo and standard placebo. Cochrane Database Syst Rev. 2023 Mar 6;3(3):MR000055. doi: 10.1002/14651858.MR000055.pub2. PMID 36877132